CLINICAL TRIAL: NCT00222222
Title: Mediators of Inflammation, Prognostic Markers and Genetic Polymorphisms in Patients With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Dr. med. Ursula Hoffmann, PD Dr. med., Universitätsmedizin Mannheim
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Nr.0244.4_1; 0244.4
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Sepsis
Keywords: severe sepsis; prognostic markers; polymorphisms; SIRS
MeSH Terms: conditions — Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: vein puncture — comparison of different inflammatory markers in the blood of septic patients

SUMMARY:
Aims of the study were to find vascular markers of inflammation and endothelial damage during the course of severe sepsis in septic patients and the effects of treatment with anti-inflammatory medication (such as Drotregocin alfa (activated)). Another aim is to find new markers and gene polymorphisms for prognosis and mortality of patients with severe sepsis. The hypothesis is that higher plasma concentrations of certain markers in septic patients are associated with a higher mortality rate.

DETAILED DESCRIPTION:
During the past years many investigators have focused on the immunological changes in sepsis disease, and great attention has been paid to the development of practicable means of immunomonitoring. Human activated protein C (Drotrecogin alfa (activated)), an important coagulation inhibitor plays a major role in regulating microvascular coagulation, inflammation and immunology. Little is known about prognostic vascular biomarkers during the time course of patients with severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* SIRS-Criteria
* Proven Infection
* One sepsis-induced organ-failure
* Adults <18 years old

Exclusion Criteria:

* Anemia
* Pregnancy
* Blood donor in the last 3 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2003-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
New Prognostic markers for septic patients | until 300 Patients are included

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Hoffmann, MD, Principal Investigator — First Department of Medicine, University Medical Centre Mannheim; Michael Behnes, MD, Study Chair — University Medical Centre Mannheim
Locations (1):
- 1. Medical Department, University Hospital Mannheim, Mannheim, Germany

REFERENCES:
- [Derived] Behnes M, Brueckmann M, Lang S, Putensen C, Saur J, Borggrefe M, Hoffmann U. Alterations of leptin in the course of inflammation and severe sepsis. BMC Infect Dis. 2012 Sep 14;12:217. doi: 10.1186/1471-2334-12-217. PMID 22973876